CLINICAL TRIAL: NCT01917084
Title: Training in Exercise Activities and Motion for Growth (A Study Conducted by the Pediatric Heart Network)
Brief Title: Training in Exercise Activities and Motion for Growth
Acronym: T4G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: U10HL068270 (NIH); U01HL068270 (NIH)
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Results first posted 2021-01-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2013-12

CONDITIONS: Single Ventricle Physiology
Keywords: Passive range of motion; Single ventricle; Infants; Congenital heart disease
MeSH Terms: conditions — Univentricular Heart; Heart Defects, Congenital | interventions — Range of Motion, Articular; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Passive range of motion (ROM) exercise (Experimental): A 10 - 15 minute passive range of motion (ROM) exercise program will be administered daily during hospitalization for up to 21 days or until discharge (whichever comes first).
  Interventions: Other: Passive range of motion (ROM) exercise

INTERVENTIONS:
Other: Passive range of motion (ROM) exercise — After their Norwood surgery, stable subjects will undergo passive ROM exercise therapy for up to 21 consecutive days or until hospital discharge, whichever comes first. Subjects will have completed the study after their anthropometric measurements are collected at 3 months of age

SUMMARY:
To determine if an exercise program of passive range of motion (ROM) is safe and feasible in infants with single ventricle (SV) physiology after their Norwood procedure.

DETAILED DESCRIPTION:
This is a non-randomized pilot study to evaluate the safety and feasibility of an exercise program in hospitalized infants with single ventricle physiology. Following the Norwood procedure, the intervention will be administered for up to 21 days or until discharge, whichever comes first. Data will be collected daily during hospitalization and at a follow-up visit at 3 months of age. Sources of data will include medical record review. Twenty subjects will be enrolled at three Pediatric Heart Network study sites (Utah Primary Children's Hospital, Children's Hospital of Philadelphia and Texas Children's Hospital). Subjects will be recruited following Institutional Review Board (IRB) approval at each institution and parental/legal guardian consent.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized infants with SV physiology
* >37 weeks gestation
* <30 days of age
* Hemodynamically stable (as defined by the attending physician) after surgical or interventional palliation with closed sternum
* Parent or guardian willing to comply with protocol and provide written informed consent

Exclusion Criteria:

* Intrauterine growth restriction
* Chromosomal or recognizable phenotypic syndrome of non-cardiac congenital abnormalities associated with growth failure (for example Trisomy, Noonan or Turner syndromes)
* Unstable hemodynamics as defined by the attending physician
* Non-cardiac diagnosis associated with growth failure
* Severe neurologic injury resulting from stroke or intracranial hemorrhage confirmed by head CT/ MRI or cranial ultrasound
* Anticipated discharge within 14 days of screening

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Lambert, MSN, c-FNP, Study Chair — Utah Primary Children's Medical Center
Locations (3):
- United States (3):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine - Texas Children's Hospital, Houston, Texas
  - Utah Primary Children's Medical Center, Salt Lake City, Utah

REFERENCES:
- See also: Pediatric Heart Network — https://www.pediatricheartnetwork.org/studies/passive-range-of-motion-team-4-growth/

RESULTS

PARTICIPANT FLOW:
Groups:
- Passive Range of Motion (ROM) Exercise: A 10 - 15 minute passive range of motion (ROM) exercise program was administered daily during hospitalization for up to 21 days or until discharge (whichever came first).
  Passive range of motion (ROM) exercise: After their Norwood surgery, stable subjects underwent passive ROM exercise therapy for up to 21 consecutive days or until hospital discharge, whichever came first. Subjects completed the study after their anthropometric measurements were collected at 3 months of age
Period: Overall Study
Arm/Group | Passive Range of Motion (ROM) Exercise
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Passive Range of Motion (ROM) Exercise
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: days] | 8 [5 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AEs) and Serious Adverse Events (SAEs) in a Passive ROM Exercise Program, Administered up to 21 Days After the Norwood Procedure, in Infants With Single Ventricle Physiology
Description: * Number of adverse events (AE), of any type, occurring during and for one hour after the daily study intervention is concluded
  * Number of AEs that are possibly or probably related to the intervention occurring during and for one hour after the daily study intervention is concluded
  * Number of Serious Adverse Events (SAEs) possibly or probably related to the intervention occurring at any time during the 21 day intervention period
Time Frame: during the intervention and for one hour afterwards, daily up to 21 days
Measure: Number; unit: events
Arm/Group | Passive Range of Motion (ROM) Exercise
Number analyzed (Participants) | 20
events
  Number of adverse events | 11
  Number of AEs that are possibly or probably relate | 1
  Number of SAEs possibly or probably related | 0

2. Primary Outcome: Feasibility of a Passive ROM Exercise Program, Administered up to 21 Days After the Norwood Procedure, in Infants With Single Ventricle Physiology
Description: Percentage of days with high completion, medium completion, and low completion of the intervention:
  * High completion is defined as >75% of the intervention
  * Medium completion is defined as 50-75% of the intervention
  * Low completion is defined as <50% of the intervention
  Percentage of days with high/medium/low completion was then calculated across all participants and days
Time Frame: during intervention, up to 21 days
Measure: Number; unit: percent of days
Arm/Group | Passive Range of Motion (ROM) Exercise
Number analyzed (Participants) | 20
percent of days
  High completion | 88
  Medium completion | 2
  Low completion | 10

3. Primary Outcome: Number of Participants With Adverse Events (AEs) in a Passive ROM Exercise Program, Administered up to 21 Days After the Norwood Procedure, in Infants With Single Ventricle Physiology
Description: • Number of participants with adverse events (AE), of any type, occurring during and for one hour after the daily study intervention is concluded
Time Frame: during the intervention and for one hour afterwards, daily up to 21 days
Measure: Number; unit: participants
Arm/Group | Passive Range of Motion (ROM) Exercise
Number analyzed (Participants) | 20
participants | 6

ADVERSE EVENTS:
Time Frame: through final (pre-Stage II palliation) study visit, which occurred at a different age and time from initial surgery for each participant, typically at 3-6 months of age
Arm/Group | Passive Range of Motion (ROM) Exercise
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Passive Range of Motion (ROM) Exercise (N=20)
cardiac arrest (Cardiac disorders) | 1 (1)
hypercarbia secondary to oversedation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
laryngomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
respiratory distress with hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Passive Range of Motion (ROM) Exercise (N=20)
Intermittent Sinus Tachycardia (Cardiac disorders) | 1 (1)
Poor weight gain (General disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachypnic with feeds (Respiratory, thoracic and mediastinal disorders) | 1 (1)
increased work of breathing with feeds (Respiratory, thoracic and mediastinal disorders) | 1 (1)
midsternal wound dehiscence (Skin and subcutaneous tissue disorders) | 1 (1)
ventricular bigeminy (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No